CLINICAL TRIAL: NCT07400419
Title: Effects of Resistance Exercise Among TGD Individuals Initiating Estrogen-Based Gender-Affirming Hormone Therapy
Acronym: STRENGTH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Mabel Toribio, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025P003023
Record Dates: First submitted 2026-01-28; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Muscle Mass and Strength
Keywords: Transgender women; Gender-Diverse; Estrogen-dominant gender-affirming hormone therapy; Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance Exercise Intervention (Active Comparator): Participants in this arm will be randomized to a 12-week at-home resistance exercise program.
  Interventions: Behavioral: Resistance Exercise Program; Behavioral: Nutrition and Exercise Counseling
- No exercise intervention (Placebo Comparator): Participants in this arm will receive educational counseling on nutrition and exercising.
  Interventions: Behavioral: Nutrition and Exercise Counseling

INTERVENTIONS:
Behavioral: Resistance Exercise Program — Participants will initiate this program at the time that they start their gender-affirming hormone therapy and will be instructed to complete resistance exercises for three 60-minute sessions per week for 12 weeks. Participants will have a weekly video call to demonstrate the exercises for that week, have a supervised training session to ensure exercises are performed safely and as instructed, monitor their continued participation in the exercise intervention, and answer any questions or issues that arise as part of the program. Further, participants will be provided with resistance bands, a TRX suspension trainer, and dumbbell weights in order to complete the resistance exercises for the program. Examples of how each exercise can be modified depending on a participant's limitations will also be provided as needed. The study team will ascertain whether they can progress to the next week's exercises depending on their ability to achieve the number of repetition's of the prior week.
  Arms: Resistance Exercise Intervention
Behavioral: Nutrition and Exercise Counseling — Participants will undergo lifestyle counseling related to optimization of their nutrition and exercise regimen.

SUMMARY:
Estrogen-dominant gender-affirming hormone therapy (GAHT) is standard of care for transgender women and gender-diverse individuals and typically consists of estrogen together with anti-androgen/ testosterone therapy. Estrogen and testosterone balance influences fat and muscle mass, muscular strength and the development of sarcopenia. Sarcopenia, a condition characterized by the loss of muscular mass, strength, and function, in turn, is associated with increased mortality and adverse health outcomes. Estrogen-dominant GAHT may have deleterious effects on body composition and muscular performance that place TGD individuals at-risk for sarcopenia. As part of NCT04128488, our investigative team found that appendicular lean mass (ALM)/ height2 decreases after estrogen-based GAHT, thereby portending a higher risk for sarcopenia after GAHT. Early recognition of the changes in body composition and muscular performance leading to sarcopenia are critical, providing potential avenues to intervene and abrogate untoward downstream health effects. A promising intervention is resistance exercise, which has been shown in select populations to improve muscular mass and strength and reduce fat mass, and, thus, mitigate progression to sarcopenia in at-risk populations. For this prospective, pilot clinical trial, investigators will enroll participants who are about to be initiated on estrogen-dominant gender-affirming hormone therapy. Investigators will be randomizing participants 1:1 to either an at-home resistance exercise intervention or no exercise intervention (nutritional and exercise counseling only) for 12 weeks and assess muscle mass, strength, and function both before and after this 12-week period. The exercise intervention group will be provided with the necessary materials to complete the exercise program along with weekly virtual visits with our study team in order to learn their assigned exercises for the week. Further, survey tools will be administered to ascertain whether the resistance exercise intervention may affect gender congruence.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Initiating GAHT with estradiol (oral, sublingual, patch, injection) AND androgen suppression (leuprolide, spironolactone or bicalutamide)
* Identifies as either a transgender female/woman, gender-diverse, non-binary, gender non-confirming, gender-fluid, and/or gender-queer
* Assigned male sex at birth

Exclusion Criteria:

* Current condition(s) which may preclude the ability to participate in a resistance exercise program (including but not limited to conditions which may significantly impair mobility and balance)
* Current condition(s) where resistance exercise program may be contraindicated (including but not limited to decompensated heart failure, unstable ischemic heart disease, pulmonary hypertension, aortic aneurysm, moderate to severe valvopathies, and/or moderate to severe chronic respiratory insufficiency)
* Use of testosterone therapy for > 1 month in the last 6 months
* Use of gender-affirming hormone therapy with androgen/testosterone suppression and/or estradiol therapy within 1 year of enrollment
* Use of gender-affirming hormone therapy with androgen/testosterone suppression and/or estradiol therapy for > 1 year at any time period prior to enrollment
* History of an orchiectomy
* Current resistance exercise (including but not limited to use of resistance bands, suspension equipment, body weight exercise, free weight exercise) of 60 minutes or greater per week
* Enrollment in another study that the study investigators deem as potentially interfering with study participants or study endpoints

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender female/woman, gender-diverse, non-binary, gender non-confirming, gender-fluid, and/or gender-queer
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Appendicular lean mass/height^2 | 12 weeks
  Change in appendicular lean mass/height^2 (kg/m^2) assessed via whole body DEXA in resistance exercise group
Gender congruence | 12 weeks
  Change in gender congruence (utilizing the total scale score from Transgender Congruence Scale) in resistance exercise group

SECONDARY OUTCOMES:
Visceral adipose tissue mass | 12 weeks
  Change in total visceral adipose tissue mass (g) assessed using whole body DEXA in resistance exercise group
Visceral adipose tissue volume | 12 weeks
  Change it total visceral adipose tissue volume (cm3) assessed using whole body DEXA in resistance exercise group
Total fat mass | 12 weeks
  Change in total fat mass (kg) assessed using whole body DEXA in resistance exercise group
Total lean body mass | 12 weeks
  Change in total lean body mass (kg) assessed using whole body DEXA in resistance exercise group
Muscular function | 12 weeks
  Change in muscular function assessed via the 5 X sit to stand test (sec) in resistance exercise group
Hand-grip strength | 12 weeks
  Change in hand-grip strength (kg) assessed using a Lafayette Hand Grip Dynamometer in resistance exercise group
Horizontal shoulder adduction strength | 12 weeks
  Change in horizontal shoulder adduction strength (kgf) assessed using a Hogan Scientific MicroFET2 Handheld dynamometer in resistance exercise group
Shoulder extension strength | 12 weeks
  Change in shoulder extension strength (kgf) assessed using a Hogan Scientific MicroFET2 Handheld dynamometer in resistance exercise group
Elbow flexion strength | 12 weeks
  Change in elbow flexion strength (kgf) assessed using a Hogan Scientific MicroFET2 Handheld dynamometer in resistance exercise group
Elbow extension strength | 12 weeks
  Change in elbow extension strength (kgf) assessed using a Hogan Scientific MicroFET2 Handheld dynamometer in resistance exercise group
Knee extension strength | 12 weeks
  Change in knee extension strength (kgf) assessed using a Hogan Scientific MicroFET2 Handheld dynamometer in resistance exercise group
Knee flexion strength | 12 weeks
  Change in knee flexion strength (kgf) assessed using a Hogan Scientific MicroFET2 Handheld dynamometer in resistance exercise group
Hip extension strength | 12 weeks
  Change in hip extension strength (kgf) assessed using a Hogan Scientific MicroFET2 Handheld dynamometer in resistance exercise group
Resting energy expenditure | 12 weeks
  Change in resting energy expenditure (kcal/day) assessed using a metabolic cart in the resistance exercise group
Resting metabolic rate | 12 weeks
  Change in resting metabolic rate (kcal/day) assessed using a metabolic cart in resistance exercise group
Respiratory quotient | 12 weeks
  Change in respiratory quotient (ratio) assessed using a metabolic cart in the resistance exercise group
Between-group change in appendicular lean body mass/ height^2 | 12 weeks
  Between-group change in appendicular lean body mass/ height^2 (kg/m^2) assessed via whole body DEXA
Between-group change in total visceral adipose tissue mass | 12 weeks
  Between-group change in total visceral adipose tissue mass (g) assessed using whole body DEXA
Between-group change in visceral adipose tissue volume | 12 weeks
  Between-change in total visceral adipose tissue volume (cm3) assessed using whole body DEXA
Between-group change in total fat mass | 12 weeks
  Between-change in total fat mass (kg) assessed using whole body DEXA
Between-group change in total lean body mass | 12 weeks
  Between-group change in total lean body mass (kg) assessed using whole body DEXA
Between-group change in muscular function via the 5x sit to stand test | 12 weeks
  Between-group change in muscular function assessed via the 5 X sit to stand test (sec)
Between-group change in hand-grip strength | 12 weeks
  Between-group change in hand-grip strength (kg) assessed using a Lafayette Hand Grip Dynamometer
Between-group change in horizontal shoulder adduction strength | 12 weeks
  Between-group change in horizontal shoulder adduction strength (kgf) assessed using a Hogan Scientific MicroFET2 Handheld dynamometer
Bwtween-group change in shoulder extension strength | 12 weeks
  Between-group change in shoulder extension strength (kgf) assessed using a Hogan Scientific MicroFET2 Handheld dynamometer
Between-group change in elbow flexion strength | 12 weeks
  Between-group change in elbow flexion strength (kgf) assessed using a Hogan Scientific MicroFET2 Handheld dynamometer
Between-group change in elbow extension strength | 12 weeks
  Between-group change in elbow extension strength (kgf) assessed using a Hogan Scientific MicroFET2 Handheld dynamometer
Between-group change in knee extension strength | 12 weeks
  Between-group change in knee extension strength (kgf) assessed using a Hogan Scientific MicroFET2 Handheld dynamometer
Between-group change in knee flexion strength | 12 weeks
  Between-group change in knee flexion strength (kgf) assessed using a Hogan Scientific MicroFET2 Handheld dynamometer
Between-group change in hip extension strength | 12 weeks
  Between-group change in hip extension strength (kgf) assessed using a Hogan Scientific MicroFET2 Handheld dynamometer
Between-group change in resting energy expenditure | 12 weeks
  Between-group change in resting energy expenditure (kcal/day) assessed using a metabolic cart
Between-group change in resting metabolic rate | 12 weeks
  Between-group change in resting metabolic rate (kcal/day) assessed using a metabolic cart
Between-group change in respiratory quotient | 12 weeks
  Between-group change in respiratory quotient (ratio) assessed using a metabolic cart
Appearance congruence | 12 weeks
  Change in appearance congruence (utilizing the appearance congruence subscale score from Transgender Congruence Scale) in resistance exercise group
Gender identity acceptance | 12 weeks
  Change in gender identity acceptance (utilizing the gender identity acceptance subscale score from Transgender Congruence Scale) in resistance exercise group
Between-group change in appearance congruence | 12 weeks
  Between-group change in appearance congruence (utilizing the appearance congruence subscale score from Transgender Congruence Scale)
Between-group change in gender identity acceptance | 12 weeks
  Between-group change in gender identity acceptance (utilizing the gender identity acceptance subscale score from Transgender Congruence Scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided